CLINICAL TRIAL: NCT07242625
Title: A Multi-center, Prospective, Compared, Randomized, Evaluator-blinded, Pilot Study to Evaluate the Effectiveness of Digital Therapeutics 'NDTx-02' on Executive Function in Children and Adolescents With Attention-Deficit/Hyperactivity Disorder (ADHD) or Autism Spectrum Disorder (ASD)
Brief Title: A Pilot Study on Efficacy of Digital Therapeutic NDTx-02 for Executive Function in Children and Adolescents With ADHD or ASD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neudive Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ND-05; DIP2024BrainAI (Other Grant/Funding Number: Daegu Digital Innovation Promotion Agency (DIP))
Record Dates: First submitted 2025-09-29; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Attention-Deficit/Hyperactivity Disorder; Autism Spectrum Disorder
Keywords: Attention-Deficit/Hyperactivity Disorder; Autism Spectrum Disorder; Digital therapeutics; Executive function; Children; Adolescents; Self-management skills; Cognitive Behavior Therapy; Intervention
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (immediate intervention) (Experimental): NDTx-02 + TAU for the first 6 weeks (stage 1), followed by TAU only for the following 6 weeks (stage 2).
  Interventions: Device: NDTx-02 + TAU; Behavioral: TAU
- The waitlist control group (delayed intervention) (Other): TAU only during the first 6 weeks (stage 1), followed by NDTx-02 + TAU for the following 6 weeks (stage 2).
  Interventions: Behavioral: TAU

INTERVENTIONS:
Device: NDTx-02 + TAU — NDTx-02 intervention: Participants will be provided with a tablet pre-installed with NDTx-02 and instructed to use the device five times per week for six weeks, for a total of 30 sessions.
  Arms: The experimental group (immediate intervention)
Behavioral: TAU — TAU (Treatment-As-Usual): Attention-Deficit/Hyperactivity Disorder (ADHD) or Autism Spectrum Disorder (ASD)-related treatment/rehabilitation/education.

SUMMARY:
The purpose of this study is to explore the preliminary safety and effectiveness of the digital therapeutic device 'NDTx-02' in supporting improvements of executive function in children and adolescents diagnosed with Attention-Deficit/Hyperactivity Disorder (ADHD) or Autism Spectrum Disorder (ASD).

DETAILED DESCRIPTION:
This pilot clinical trial aims to evaluate the preliminary safety and effectiveness of NDTx-02 in combination with Treatment-As-Usual (TAU) compared with TAU alone (waitlist control).

The study will employ a randomized waitlist-control design, in which participants will be assigned to either experimental group (immediate intervention) or waitlist control group (delayed intervention) with a 1:1 ratio.

* Experimental group (immediate intervention): NDTx-02 + TAU for the first 6 weeks (stage 1), followed by TAU only for the following 6 weeks (stage 2).
* Waitlist control group (delayed intervention): TAU only during the first 6 weeks (stage 1), followed by NDTx-02 + TAU for the following 6 weeks (stage 2).

Efficacy will be assessed using the K-BRIEF-2, K-VABS-II, K-ARS-5, KAT, WMT, C-TMT, Stroop Color and Word Test Children's Version, Digit Span test, CGI-S, and CGI-I.

The primary efficacy analysis will compare the experimental group and the waitlist control group during Stage 1 (weeks 0-6). The delayed intervention period (Stage 2) will be analyzed as secondary/exploratory.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 5 to 12 years at the time of screening
* Diagnosed with Attention-Deficit/Hyperactivity Disorder (ADHD) or Autism Spectrum Disorder (ASD)* by a psychiatrist according to DSM-5 diagnostic criteria

  *For ASD, diagnosis can be supported by the Autism Diagnostic Interview-Revised (ADI-R) or the Autism Diagnostic Observation Schedule (ADOS), either version 1 or 2
* Full-Scale Intelligence Quotient (FSIQ) of 65 or higher
* Able to use the 'NDTx-02' installed on a tablet, alone or with the assistance of a guardian
* Able to comply with the recommended application schedule for the investigational device (6 weeks, 30 sessions, 5 times per week)
* Agree not to add or change any treatment/education/rehabilitation programs or medications, including Applied Behavior Analysis (ABA) or cognitive therapy, during the study period (continuation of pre-existing TAU [Treatment-As-Usual] is allowed)
* Participant and parent (or legal guardian) voluntarily decide to join the trial and provide written informed consent
* Participants willing to comply with the clinical trial procedures

Exclusion Criteria:

* A risk of clinically significant behavioral problems, emotion regulation problems, psychotic symptoms, self-harm, or other harm at a level that affects the treatment process
* Severe acute/chronic medical or mental illness
* Serious trauma or surgery performed within 4 weeks before the screening date
* Participants with other disabilities such as severe neurological diseases (e.g. brain lesions, mental disorders, etc.)
* Participants who are currently participating in another clinical trial or have participated in another clinical trial within 30 days before the screening date
* Change in the dosage or regimen of medications that may significantly affect cognitive function within 4 weeks prior to the baseline visit
* Change in participation in treatment/education/rehabilitation programs that may significantly affect cognitive function within 4 weeks prior to the baseline visit
* Participation in a clinical trial of, or prior experience using, cognitive improvement or daily living improvement software within 12 weeks prior to the baseline visit
* In other cases where the investigator determines that participation in the clinical trial is inappropriate due to ethical reasons or the possibility of influencing the results of the clinical trial

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
K-BRIEF-2 (Behavior Rating Inventory of Executive Function, Second Edition) | Baseline (V2,V4), Day 42 (V4,V6)
  The K-BRIEF-2 consists of 63 items rated on a 3-point scale (Never, Sometimes, Often). The K-BRIEF-2 comprises 9 scales (Inhibit, Self-Monitor, Shift, Emotional Control, Initiate, Working Memory, Plan/Organize, Task-Monitor, Organization of Materials) organized under 3 index scores (Behavior Regulation, Emotion Regulation, Cognitive Regulation). The 9 scales collectively yield the Global Executive Composite (GEC), which reflects overall executive functioning. Higher T scores indicate greater executive function difficulties.

SECONDARY OUTCOMES:
K-ARS-5 (Korean ADHD Rating Scale, 5th Edition) | Baseline (V2,V4), Day 42 (V4,V6)
  The K-ARS-5 is a parent-rated scale for children aged 5-12, developed based on DSM-5 diagnostic criteria for ADHD. It contains 30 items that assess the frequency and severity of ADHD symptoms, including inattention and hyperactivity/impulsivity. Higher scores indicate greater ADHD symptom severity.
K-VABS-II (Korean Vineland Adaptive Behavior Scales-II) | Baseline (V2,V4), Day 42 (V4,V6)
  The K-VABS-II is a clinician-administered tool for individuals from 0 to 99 years of age, assessing social and adaptive functioning across Communication, Daily Living Skills, Socialization, and Motor Skills, as well as a Maladaptive Behavior Index. It consists of 433 items. Standard scores range from 55 to 145, with higher scores reflecting better adaptive functioning.
KAT (Korean Attention Test System) | Baseline (V2,V4), Day 42 (V4,V6)
  The KAT is an assessment tool for children aged 5-15 that systematically evaluates visual and auditory attention. It provides measures such as omission errors, commission errors, mean reaction time, and ADHD indices, and is designed to identify attention deficits and impulsivity.
WMT (Working Memory Test for Children) | Baseline (V2,V4), Day 42 (V4,V6)
  The WMT is an assessment tool for children aged 5-15, designed to measure working memory capacity. It evaluates performance in forward and backward sequencing tasks, as well as longest span achieved. Scores provide insight into attention and working memory deficits, particularly for ADHD diagnosis.
C-TMT (Color Trail Making Test for Children) | Baseline (V2,V4), Day 42 (V4,V6)
  The C-TMT is an assessment tool for children aged 5-15 that measures executive function and cognitive flexibility. It assesses completion times, sequencing errors, and interference indices. Poorer performance (longer completion time, more errors) indicates executive dysfunction, often associated with ADHD.
Stroop Color and Word Test - Children's Version | Baseline (V2,V4), Day 42 (V4,V6)
  The Stroop Children's Test assesses frontal lobe function and inhibitory control in children aged 5-14. It evaluates words, color, color-word, and interference scores. It is used in the diagnosis of ADHD, tic disorders, learning disabilities, and autism spectrum disorder, as well as in assessing neuropsychological deficits.
Digit Span Test | Baseline (V2,V4), Day 42 (V4,V6)
  The Digit Span subtest of the K-WISC-V assesses auditory attention and working memory. It includes Digit Span Forward, Digit Span Backward, and Digit Span Sequencing, as well as the longest span achieved in each category. Higher scores indicate better memory capacity and attentional control.
CGI-S (Clinical Global Impression-Severity) | Baseline (V2,V4), Day 42 (V4,V6)
  The CGI-S is a clinician-rated scale assessing overall illness severity on a 7-point scale (1 = normal, 7 = extremely severe). Clinicians rate current severity relative to past patients with the same diagnosis, providing a standardized severity assessment.
CGI-I (Clinical Global Impression-Improvement) | Day 42 (V4,V6)
  The CGI-I is a clinician-rated scale assessing overall improvement or worsening of the patient's condition compared to baseline. It is rated on a 7-point scale (1 = very much improved, 7 = very much worse). Lower scores indicate greater clinical improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Yoo-Sook Joung, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (3):
- South Korea (3):
  - Daegu Catholic University Medical Center, Daegu
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No